CLINICAL TRIAL: NCT00893971
Title: A Randomized, Double-blind, Single Dose, Four-period, Four-treatment, Cross-over Study Evaluating the Safety of PT001, PT003, PT005 Administered Individually and PT001 + PT005 Delivered Together in Separate Inhalers in Healthy Subjects
Brief Title: Study to Evaluate Single Inhaled Doses of PT001, PT003, PT005 and PT001 Plus PT005 in Healthy Subjects
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Pearl Therapeutics, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Quadruple | Purpose: Treatment
Other Study IDs: PT0030901
Record Dates: First submitted 2009-05-05; First posted 2009-05-06 (Estimated); Results first posted 2017-04-26 (Actual); Last update posted 2017-04-26 (Actual); Status verified 2017-03

CONDITIONS: Healthy Volunteers
Keywords: Healthy Volunteers

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (4):
- 1 (Experimental): Inhaled PT001 18 μg
  Interventions: Drug: PT001
- 2 (Experimental): Inhaled PT005 2.4 μg
  Interventions: Drug: PT005
- 3 (Experimental): Inhaled PT003 (PT001 18 μg / 2.4 μg PT005)
  Interventions: Drug: PT003
- 4 (Experimental): PT001 18 μg + PT005 2.4 μg
  Interventions: Drug: PT001 + PT005

INTERVENTIONS:
Drug: PT001 — Inhaled PT001, single dose
  Arms: 1
Drug: PT005 — Inhaled PT005, single dose
  Arms: 2
Drug: PT003 — Inhaled PT003, single dose
  Arms: 3
Drug: PT001 + PT005 — Inhaled PT001 + PT005, single dose
  Arms: 4

SUMMARY:
The purpose of this study is to evaluate the safety of a single dose of PT003 compared with single doses of PT001 and PT005, and compared with PT001 plus PT005 delivered together as two separate single doses in healthy subjects.

ELIGIBILITY:
Inclusion Criteria:

* Provide signed written informed consent
* 18-55 years of age
* Healthy subjects confirmed by medical history, physical examination, vital signs, pulmonary function tests, electrocardiogram and clinical laboratory tests
* Female subjects of child-bearing potential who are sexually active must be willing to undergo a pregnancy test and agree to use two forms of contraception
* Body mass index (BMI) between 18.5 and 30, inclusive
* Non-smokers for at least 6 months prior to screening
* Pulmonary function tests within normal limits
* Willing to remain at the study center for at least 12-24 hours on each test day
* Venous access in both arms to allow collection of numerous blood samples

Exclusion Criteria:

* Women who are pregnant or lactating
* Clinically significant medical conditions
* Viral illness within the last 30 days
* Symptomatic prostatic hypertrophy or bladder neck obstruction
* Known narrow-angle glaucoma
* History of bowel obstruction
* Clinically significant abnormal electrocardiogram
* Positive Hepatitis B surface antigen or positive Hepatitis C antibody
* Positive screening test for HIV antibodies
* History of hypersensitivity to any beta2-agonists, anticholinergics, or any component of the MDI
* Known or suspected history of alcohol or drug abuse within the last 2-years
* Greater than normal alcohol consumption
* Ingestion of any poppy seeds within the 48 hours prior to the screening
* Ingestion of any poppy seeds within the 48 hours prior to, or any alcohol, xanthines or grapefruit-containing foods or beverages within the 24 hours prior to, or during, each confinement
* Positive breath alcohol result
* Positive urine drug screen
* Use of any beta2-agonists,or anticholinergics prior to the recruitment interview
* Lower respiratory tract infections requiring antibiotics in the previous 6 weeks
* Use of any other prescription medication
* Use of any over the counter product, herbal product, diet aid, hormone supplement
* Donation > 450 ml of blood within 8 weeks of first treatment dose
* Clinically significant vital sign abnormality
* Clinically significant biochemical, hematological or urinalysis abnormality
* Affiliations with investigator site
* Treatment with investigational study drug or participation in another clinical trial or study within the last 30 days or 5 half lives prior to screening, whichever is longer

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 16 (Actual)
Dates: Start 2009-05; Primary Completion 2009-07 (Actual); Study Completion 2009-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Colin Reisner, M.D., Study Director — Pearl Therapeutics
Locations (1):
- Dr Joanne Marjason, Herston, Queensland, Australia

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Conducted at a single site in Australia from May 2009 through July 2009. Study participation was a maximum of 7 weeks.
Pre-assignment Details: Study evaluating a single administration of inhaled treatment (PT001, PT003, PT005 and PT001+PT005 delivered from separate inhalers as a loose combination).Each subject was randomized to 1 of 4 sequences. Each sequence included the four treatment groups.
Groups:
- Overall Study: All patients randomized
Period: Overall Study
Arm/Group | Overall Study
Started | 16
Placebo + GP MDI (PT001) | 15
Placebo + GFF MDI (PT003) | 15
Placebo + FF MDI (PT005) | 13
GP MDI (PT001) + FF MDI (PT005) | 16
Completed | 13
Not Completed | 3
Not completed — Physician Decision | 3

BASELINE CHARACTERISTICS:
Population: All randomized subjects
Groups:
- All Subjects: Any treatment arm
Arm/Group | All Subjects
Number analyzed (Participants) | 16
Age, Continuous [Mean (Standard Deviation); unit: Years] | 27.4 (10.1)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 11
  Male | 5

OUTCOME MEASURES:

1. Primary Outcome: Symptoms of Dry Mouth
Description: Number of participants reporting dry mouth at 12 hours post-dose
Time Frame: 12 hours
Population: All subjects in the Safety Population
Measure: Number; unit: Participants
Groups:
- Placebo + PT001: Placebo + Glycopyrrolate MDI 72 µg
- Placebo + PT005: Placebo + Formoterol Fumarate 9.6 µg
- PT001 + PT005: Glycopyrrolate 72 mcg + Formoterol Fumarate 9.6 µg (taken in any order)
- Placebo + PT003: Placebo + Glycopyrrolate 72 µg/ Formoterol Fumarate µg
Arm/Group | Placebo + PT001 | Placebo + PT005 | PT001 + PT005 | Placebo + PT003
Number analyzed (Participants) | 15 | 13 | 16 | 15
Participants
  Immediately pre-dose | 3 | 1 | 3 | 1
  30 minutes post-dose | 4 | 3 | 4 | 5
  1-hour post-dose | 3 | 2 | 3 | 3
  2-hours post-dose | 3 | 1 | 3 | 1
  4-hours post-dose | 1 | 1 | 3 | 0
  6-hours post-dose | 1 | 1 | 2 | NA — If no dry mouth is present up to the 2 hr time point, then no further assessments are required. If dry mouth is present, then assessments are continued until the AE is resolved.
  8-hours post-dose | 1 | 1 | 2 | NA — If no dry mouth is present up to the 2 hr time point, then no further assessments are required. If dry mouth is present, then assessments are continued until the AE is resolved.
  12-hours post-dose | 1 | 1 | 2 | NA — If no dry mouth is present up to the 2 hr time point, then no further assessments are required. If dry mouth is present, then assessments are continued until the AE is resolved.

2. Primary Outcome: Symptoms of Tremor
Description: Number of participants reporting tremor at 12 hours post-dose
Time Frame: 12 hours
Population: All subjects in the Safety Population
Measure: Number; unit: Participants
Arm/Group | Placebo + PT001 | Placebo + PT005 | PT001 + PT005 | Placebo + PT003
Number analyzed (Participants) | 15 | 13 | 16 | 15
Participants
  Immediately pre-dose | 0 | 0 | 0 | 0
  30-minutes post-dose | 0 | 0 | 0 | 0
  1-hour post-dose | 0 | 0 | 0 | 0
  2-hours post-dose | 0 | 0 | 1 | 0
  4-hours post-dose | NA — If no tremor was present at the previous 2-hour time point, no further assessment was required | 1 | 1 | NA — If no tremor was present at the previous 2-hour time point, no further assessment was required
  6-hours post-dose | NA — If no tremor was present at the previous 2-hour time point, no further assessment was required | 0 | 0 | NA — If no tremor was present at the previous 2-hour time point, no further assessment was required
  8-hours post-dose | NA — If no tremor was present at the previous 2-hour time point, no further assessment was required | NA — If no tremor was present at the previous 2-hour time point, no further assessment was required | NA — If no tremor was present at the previous 2-hour time point, no further assessment was required | NA — If no tremor was present at the previous 2-hour time point, no further assessment was required
  12-hours post-dose | NA — If no tremor was present at the previous 2-hour time point, no further assessment was required | NA — If no tremor was present at the previous 2-hour time point, no further assessment was required | NA — If no tremor was present at the previous 2-hour time point, no further assessment was required | NA — If no tremor was present at the previous 2-hour time point, no further assessment was required

3. Primary Outcome: Blood Chemistry Change From Baseline
Description: Series of 11 blood chemistries assessed throughout the study
Time Frame: 24 hours post dose for sentinel subjects, 12 hours post dose for subsequent subjects
Population: All patients in the Safety Population that had a valid measurement for the parameter
Measure: Mean (Full Range); unit: mmol/L
Arm/Group | Placebo + PT001 | Placebo + PT005 | PT001 + PT005 | Placebo + PT003
Number analyzed (Participants) | 15 | 13 | 16 | 15
mmol/L
  Sodium | 0.76 [-3 to 4] | 0.78 [-1 to 3] | 0.35 [-2 to 6] | 0.6 [-2 to 3]
  Chloride | -1.29 [-7 to 2] | -0.4 [-4 to 4] | -0.75 [-5 to 6] | -1.2 [-3 to 0]
  Urea | 0.12 [-0.9 to 1.4] | -0.05 [-1.3 to 1.8] | -0.11 [-2.6 to 1.5] | -0.33 [-3.3 to 1.1]
  Calcium | -0.01 [-0.1 to 0.08] | -0.04 [-0.2 to 0.06] | -0.03 [-0.21 to 0.08] | -0.01 [-0.11 to 0.09]
  Bicarbonate | 0.64 [-2 to 4] | 0.05 [-4 to 2] | 0.44 [-5 to 6] | 0.47 [-5 to 3]
  Glucose | -0.17 [-2.5 to 1.1] | -0.34 [-2.4 to 1.2] | -0.34 [-2 to 1.1] | 0.45 [-1.9 to 2.5]

4. Primary Outcome: Blood Chemistry Change From Baseline
Description: Series of 11 blood chemistries assessed throughout the study
Time Frame: 24 hours post dose for sentinel subjects, 12 hours post dose for subsequent subjects
Population: All subjects in the Safety Population that had a valid measurement for the parameter
Measure: Mean (Full Range); unit: µmol/L
Arm/Group | Placebo + PT001 | Placebo + PT005 | PT001 + PT005 | Placebo + PT003
Number analyzed (Participants) | 15 | 13 | 16 | 15
µmol/L
  Creatinine | 2.19 [-11 to 11] | 1.45 [-15 to 12] | 0.44 [-14 to 11] | -0.8 [-13 to 11]
  Bilirubin | -1.4 [-6 to 3] | -2.18 [-5 to 0] | -2.32 [-6 to 1] | -2.07 [-10 to 2]

5. Primary Outcome: Blood Chemistry Change From Baseline
Description: Series of 11 blood chemistries assessed throughout the study
Time Frame: 24 hours post dose for sentinel subjects, 12 hours post dose for subsequent subjects
Population: All patients in the Safety Population that had a valid measurement for the parameter
Measure: Mean (Full Range); unit: U/L
Arm/Group | Placebo + PT001 | Placebo + PT005 | PT001 + PT005 | Placebo + PT003
Number analyzed (Participants) | 15 | 13 | 16 | 15
U/L
  ALP | 2.99 [-3 to 10] | 3.59 [-3 to 12] | 1.39 [-9 to 9] | 2 [-9 to 11]
  ALT | 0.07 [-6 to 5] | -1.21 [-8 to 4] | -0.41 [-5 to 5] | -0.33 [-5 to 6]
  AST | -0.83 [-10 to 7] | 0.25 [-5 to 6] | -2.91 [-14 to 4] | -1.67 [-10 to 4]

6. Primary Outcome: Hematology Change From Baseline
Description: Hematology assessments taken throughout the study Hematocrit
Time Frame: 24 hours post dose for sentinel subjects, 12 hours post dose for subsequent subjects
Population: All subjects in the Safety Population that had a valid measurement for the parameter
Measure: Mean (Full Range); unit: % of Red Blood Cells in the blood
Arm/Group | Placebo + PT001 | Placebo + PT005 | PT001 + PT005 | Placebo + PT003
Number analyzed (Participants) | 15 | 13 | 15 | 15
% of Red Blood Cells in the blood | 0.01 [-0.07 to 0.03] | 0.01 [-0.02 to 0.04] | 0.01 [-0.02 to 0.03] | 0.01 [-0.02 to 0.04]

7. Primary Outcome: Hematology Change From Baseline
Description: Hematology assessments taken throughout the study
Time Frame: 24 hours post dose for sentinel subjects, 12 hours post dose for subsequent subjects
Population: All subjects in the Safety Population that had a valid measurement for the parameter
Measure: Mean (Full Range); unit: (10^9 cells/L)
Arm/Group | Placebo + PT001 | Placebo + PT005 | PT001 + PT005 | Placebo + PT003
Number analyzed (Participants) | 15 | 13 | 15 | 15
(10^9 cells/L)
  WCC | 17.93 [-13 to 39] | 20.61 [-1 to 55] | 10.8 [-31 to 43] | 20.33 [-17 to 54]
  Platelets | 1.08 [-1 to 3] | 0.88 [-1 to 3] | 0.93 [0 to 3] | 0.67 [-4 to 3]

8. Primary Outcome: Hematology Change From Baseline
Description: Hematology assessments taken throughout the study Hemoglobin
Time Frame: 24 hours post dose for sentinel subjects, 12 hours post dose for subsequent subjects
Population: All subjects in the Safety Population that had a valid measurement for the parameter
Measure: Mean (Full Range); unit: g/L
Arm/Group | Placebo + PT001 | Placebo + PT005 | PT001 + PT005 | Placebo + PT003
Number analyzed (Participants) | 15 | 13 | 15 | 15
g/L | 2.45 [-24 to 11] | 2.95 [-6 to 10] | 1.73 [-4 to 10] | 3.33 [-9 to 9]

9. Primary Outcome: Heart Rate Change From Baseline
Description: Change from baseline for heart rate 12-hours post-dose Heart rate (bpm)
Time Frame: 12 hours
Population: All subjects in the Safety Population that had a valid measurement for the parameter
Measure: Mean (Full Range); unit: bpm
Arm/Group | Placebo + PT001 | Placebo + PT005 | PT001 + PT005 | Placebo + PT003
Number analyzed (Participants) | 15 | 13 | 16 | 15
bpm | 2.0 [-7 to 13] | 4.4 [-12 to 21] | 2.9 [-3 to 11] | 1.8 [-13 to 19]

10. Primary Outcome: Vital Sign Change Baseline; Blood Pressure
Description: Vital sign change baseline; blood pressure
Time Frame: 12 hours
Population: All subjects in the Safety Population that had a valid measurement for the parameter
Measure: Mean (Full Range); unit: mmHg
Arm/Group | Placebo + PT001 | Placebo + PT005 | PT001 + PT005 | Placebo + PT003
Number analyzed (Participants) | 15 | 13 | 16 | 15
mmHg
  Systolic blood pressure (mmHg) | 3.3 [-14 to 18] | 1.0 [-20 to 14] | 0.1 [-9 to 14] | 0.4 [-8 to 13]
  Diastolic blood pressure (mmHg) | 6.3 [-8 to 24] | 1.5 [-13 to 10] | 0.6 [-12 to 12] | 1.6 [-14 to 28]

11. Primary Outcome: Vital Sign Change From Baseline, SpO2
Description: Vital Sign Change from baseline 12-hours post-dose SpO2 (%)
Time Frame: 12 hours
Population: All subjects in the Safety Population that had a valid measurement for the parameter
Measure: Mean (Full Range); unit: % blood oxygen saturation level
Arm/Group | Placebo + PT001 | Placebo + PT005 | PT001 + PT005 | Placebo + PT003
Number analyzed (Participants) | 15 | 13 | 16 | 15
% blood oxygen saturation level | 0.2 [-2 to 2] | 0.1 [-1 to 3] | -0.1 [-2 to 1] | 0.1 [-1 to 2]

12. Primary Outcome: ECG Change From Baseline
Description: Change from baseline for ECG parameters 12-hours post-dose Ventricular rate (bpm)
Time Frame: 12 hours
Population: Safety population
Measure: Mean (Full Range); unit: bpm
Arm/Group | Placebo + PT001 | Placebo + PT005 | PT001 + PT005 | Placebo + PT003
Number analyzed (Participants) | 15 | 13 | 16 | 15
bpm | 1.5 [-7 to 9] | 4.7 [-18 to 22] | 5.2 [-4 to 25] | 4.0 [-9 to 13]

13. Primary Outcome: ECG Change From Baseline
Description: Change from baseline for ECG parameters 12-hours post-dose
Time Frame: 12 hours
Population: Safety population
Measure: Mean (Full Range); unit: ms
Arm/Group | Placebo + PT001 | Placebo + PT005 | PT001 + PT005 | Placebo + PT003
Number analyzed (Participants) | 15 | 13 | 16 | 15
ms
  PR interval (ms) | -11.0 [-126 to 10] | -8.3 [-20 to 2] | -5.3 [-24 to 24] | -10.4 [-34 to 14]
  QRS duration (ms) | -3.0 [-10 to 4] | -5.4 [-18 to 10] | 0.4 [-10 to 42] | -2.0 [-12 to 10]
  QT interval (ms) | -8.6 [-32 to 4] | -9.4 [-42 to 20] | -10.1 [-60 to 16] | -12.8 [-26 to 10]
  QTcB (ms) | -3.7 [-24 to 18] | 5.3 [-36 to 41] | 5.4 [-17 to 39] | -2.1 [-26 to 31]
  QTcF (ms) | -5.1 [-25 to 12] | 0.0 [-19 to 16] | -0.1 [-23 to 21] | -5.9 [-18 to 24]

14. Primary Outcome: Spirometry Change From Baseline
Description: Change from baseline for spirometery measures 12-hours post-dose
Time Frame: 12 hours
Population: Safety population
Measure: Mean (Full Range); unit: Liters
Arm/Group | Placebo + PT001 | Placebo + PT005 | PT001 + PT005 | Placebo + PT003
Number analyzed (Participants) | 15 | 13 | 16 | 15
Liters
  FEV1 (L) | 0.260 [-0.28 to 0.49] | 0.148 [-0.53 to 0.43] | 0.202 [-0.27 to 0.71] | 0.195 [-0.33 to 0.49]
  FVC (L) | 0.145 [-0.51 to 0.47] | 0.0 [-0.82 to 0.44] | 0.082 [-0.49 to 0.53] | 0.045 [-0.64 to 0.50]

15. Primary Outcome: Spirometry Change From Baseline
Description: Change from baseline for spirometery measures 12-hours post-dose (FEV1 % predicted)
Time Frame: 12 hours
Population: Safety population
Measure: Mean (Full Range); unit: % predicted
Arm/Group | Placebo + PT001 | Placebo + PT005 | PT001 + PT005 | Placebo + PT003
Number analyzed (Participants) | 15 | 13 | 16 | 15
% predicted | 7.2 [-8 to 12] | 4.5 [-12 to 12] | 5.2 [-8 to 15] | 5.0 [-7 to 15]

16. Primary Outcome: Spirometry Change From Baseline
Description: Change from baseline for spirometery measures 12-hours post-dose FEV/FVC (%)
Time Frame: 12 hours
Population: Safety population
Measure: Mean (Full Range); unit: Ratio
Arm/Group | Placebo + PT001 | Placebo + PT005 | PT001 + PT005 | Placebo + PT003
Number analyzed (Participants) | 15 | 13 | 16 | 15
Ratio | 3.0 [-4 to 10] | 3.4 [0 to 7] | 3.2 [-4 to 9] | 3.6 [1 to 8]

17. Primary Outcome: Spirometry Change From Baseline
Description: Change from baseline for spirometery measures 12-hours post-dose PEFR (L/min)
Time Frame: 12 hours
Population: Safety population
Measure: Mean (Full Range); unit: L/min
Arm/Group | Placebo + PT001 | Placebo + PT005 | PT001 + PT005 | Placebo + PT003
Number analyzed (Participants) | 15 | 13 | 16 | 15
L/min | 40.4 [0 to 93] | 32.1 [-120 to 150] | 40.1 [-63 to 135] | 31.6 [-99 to 102]

18. Secondary Outcome: Plasma Glycopyrrolate PK Parameters
Description: Various pharmacokinetic parameters for plasma glycopyrrolate
Time Frame: Concentrations were measured at pre-dose and 2,5,15, and 30 minutes post dose as well as 1,2,4,6,8, and 12 hours post dose
Population: Subjects with an evaluable profile for this analyte
Measure: Mean (Standard Deviation); unit: h*pg/mL
Arm/Group | Placebo + PT001 | PT001 + PT005 | Placebo + PT003
Number analyzed (Participants) | 12 | 12 | 12
h*pg/mL
  AUC0-tlast (h*pg/mL) | 156.6 (76.7) [-0.28 to 0.49] | 100.1 (43.1) [-0.27 to 0.71] | 78.4 (36.2) [-0.33 to 0.49]
  AUC0-12 (h*pg/mL) | 156.7 (76.5) [-8 to 12] | 100.6 (42.4) [-8 to 15] | 80.1 (34.9) [-7 to 15]

19. Secondary Outcome: Plasma Glycopyrrolate PK Parameters AUC0-inf (h*pg/mL)
Description: Various pharmacokinetic parameters for plasma glycopyrrolate
Time Frame: as for outcome 18
Population: Subjects with an evaluable profile for this analyte
Measure: Mean (Standard Deviation); unit: h*pg/mL
Arm/Group | Placebo + PT001 | PT001 + PT005 | Placebo + PT003
Number analyzed (Participants) | 9 | 8 | 9
h*pg/mL | 172.4 (88.6) | 137.2 (55.4) | 100.8 (50.5)

20. Secondary Outcome: Plasma Glycopyrrolate PK Parameters (Tmax)
Description: Various pharmacokinetic parameters for plasma glycopyrrolate
Time Frame: as for outcome 18
Population: Subjects with an evaluable profile for this analyte
Measure: Mean (Standard Deviation); unit: h
Arm/Group | Placebo + PT001 | PT001 + PT005 | Placebo + PT003
Number analyzed (Participants) | 12 | 12 | 12
h | 0.16 (0.14) [-0.51 to 0.47] | 0.07 (0.06) [-0.49 to 0.53] | 0.06 (0.03) [-0.64 to 0.50]

21. Secondary Outcome: Plasma Glycopyrrolate PK Parameters (t1/2)
Description: Various pharmacokinetic parameters for plasma glycopyrrolate
Time Frame: as for outcome 18
Population: Subjects with an evaluable profile for this analyte
Measure: Mean (Standard Deviation); unit: h
Arm/Group | Placebo + PT001 | PT001 + PT005 | Placebo + PT003
Number analyzed (Participants) | 9 | 8 | 9
h | 5.34 (1.78) | 5.12 (1.61) | 5.12 (2.07)

22. Secondary Outcome: Plasma Glycopyrrolate PK Parameters Cmax (pg/mL)
Description: Various pharmacokinetic parameters for plasma glycopyrrolate
Time Frame: as for outcome 18
Population: Subjects with an evaluable profile for this analyte
Measure: Mean (Standard Deviation); unit: pg/mL
Arm/Group | Placebo + PT001 | PT001 + PT005 | Placebo + PT003
Number analyzed (Participants) | 12 | 12 | 12
pg/mL | 61.3 (40.9) [-4 to 10] | 77.8 (72.0) [-4 to 9] | 44.4 (18.3) [1 to 8]

23. Secondary Outcome: Plasma Glycopyrrolate PK Parameters (ke)
Description: Various pharmacokinetic parameters for plasma glycopyrrolate
Time Frame: as for outcome 18
Population: Subjects with an evaluable profile for this analyte
Measure: Mean (Standard Deviation); unit: 1/h
Arm/Group | Placebo + PT001 | PT001 + PT005 | Placebo + PT003
Number analyzed (Participants) | 9 | 8 | 9
1/h | 0.143 (0.047) | 0.147 (0.042) | 0.155 (0.059)

24. Secondary Outcome: Plasma Formoterol PK Parameters
Description: Various pharmacokinetic parameters for plasma formoterol
Time Frame: as for outcome 18
Population: Subjects with an evaluable profile for this analyte
Measure: Mean (Standard Deviation); unit: h*pg/mL
Arm/Group | Placebo + PT005 | PT001 + PT005 | Placebo + PT003
Number analyzed (Participants) | 11 | 11 | 11
h*pg/mL
  AUC0-tlast (h*pg/mL) | 47.9 (12.3) [-120 to 150] | 61.2 (16.5) [-63 to 135] | 57.9 (16.3) [-99 to 102]
  AUC0-12 (h*pg/mL) | 48.1 (12.2) | 61.2 (16.6) | 57.8 (16.2)

25. Secondary Outcome: Plasma Formoterol PK Parameters AUC0-inf (h*pg/mL)
Description: Various pharmacokinetic parameters for plasma formoterol
Time Frame: as for outcome 18
Population: Subjects with an evaluable profile for this analyte
Measure: Mean (Standard Deviation); unit: h*pg/mL
Arm/Group | Placebo + PT005 | PT001 + PT005 | Placebo + PT003
Number analyzed (Participants) | 8 | 7 | 8
h*pg/mL | 56.1 (8.3) | 76.4 (18.5) | 67.0 (12.8)

26. Secondary Outcome: Plasma Formoterol PK Parameters (Tmax)
Description: Various pharmacokinetic parameters for plasma formoterol
Time Frame: as for outcome 18
Population: Subjects with an evaluable profile for this analyte
Measure: Mean (Standard Deviation); unit: h
Arm/Group | Placebo + PT005 | PT001 + PT005 | Placebo + PT003
Number analyzed (Participants) | 11 | 11 | 11
h | 0.28 (0.31) [-120 to 150] | 0.27 (0.59) [-63 to 135] | 0.43 (0.46) [-99 to 102]

27. Secondary Outcome: Plasma Formoterol PK Parameters (t1/2)
Description: Various pharmacokinetic parameters for plasma formoterol
Time Frame: as for outcome 18
Population: Subjects with an evaluable profile for this analyte
Measure: Mean (Standard Deviation); unit: h
Arm/Group | Placebo + PT005 | PT001 + PT005 | Placebo + PT003
Number analyzed (Participants) | 8 | 7 | 8
h | 5.12 (1.10) | 5.28 (1.02) | 5.8 (1.32)

28. Secondary Outcome: Plasma Formoterol PK Parameters (Cmax)
Description: Pharmacokinetic parameters for plasma formoterol Cmax
Time Frame: as for outcome 18
Population: Subjects with an evaluable profile for this analyte
Measure: Mean (Standard Deviation); unit: pg/mL
Arm/Group | Placebo + PT005 | PT001 + PT005 | Placebo + PT003
Number analyzed (Participants) | 11 | 11 | 11
pg/mL | 10.4 (3.8) [-120 to 150] | 13.2 (4.5) [-63 to 135] | 11.9 (4.0) [-99 to 102]

29. Secondary Outcome: Plasma Formoterol PK Parameters (ke)
Description: Pharmacokinetic parameters for plasma formoterol ke
Time Frame: as for outcome 18
Population: Subjects with an evaluable profile for this analyte
Measure: Mean (Standard Deviation); unit: 1/h
Arm/Group | Placebo + PT005 | PT001 + PT005 | Placebo + PT003
Number analyzed (Participants) | 8 | 7 | 8
1/h | 0.142 (0.035) [-120 to 150] | 0.135 (0.025) [-63 to 135] | 0.126 (0.032) [-99 to 102]

30. Primary Outcome: Serum Potassium Change From Baseline
Time Frame: 12 hours
Population: All subjects in the Safety Population
Measure: Median (Full Range); unit: mmol/L
Arm/Group | Placebo + PT001 | Placebo + PT005 | PT001 + PT005 | Placebo + PT003
Number analyzed (Participants) | 14 | 12 | 15 | 14
mmol/L | 4.4 [4.0 to 5.1] | 4.1 [3.5 to 4.9] | 4.1 [3.7 to 4.8] | 4.2 [3.8 to 4.7]

ADVERSE EVENTS:
Time Frame: Adverse events and serious adverse events were collected from the time the subject signed consent until final visit or discontinuation visit.
Description: Safety population included all participants who received investigational drug; participants were included in safety population according to the investigational drug they were receiving at the time of the event.
Arm/Group | Placebo + PT001 | Placebo + PT005 | PT001 + PT005 | Placebo + PT003
Serious Adverse Events (participants affected / at risk) | 0/15 | 0/13 | 0/16 | 0/15
Other Adverse Events (participants affected / at risk) | 7/15 | 6/13 | 8/16 | 9/15
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Placebo + PT001 (N=15) | Placebo + PT005 (N=13) | PT001 + PT005 (N=16) | Placebo + PT003 (N=15)
Dry eye (Eye disorders) | 1 (1) | 1 (1) | 0 (0) | 1 (1)
Dry mouth (Gastrointestinal disorders) | 2 (2) | 3 (3) | 4 (4) | 4 (4)
Toothache (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Chest discomfort (General disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Upper respiratory tract infection (Infections and infestations) | 0 (0) | 1 (1) | 1 (1) | 1 (1)
Contusion (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Muscle tightness (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Dizziness (Nervous system disorders) | 1 (1) | 1 (1) | 1 (1) | 1 (1)
Headache (Nervous system disorders) | 2 (3) | 1 (1) | 1 (1) | 5 (5)
Tremor (Nervous system disorders) | 0 (0) | 1 (1) | 2 (2) | 1 (1)
Dysmenorrhea (Reproductive system and breast disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Rhinitis (Respiratory, thoracic and mediastinal disorders) | 2 (3) | 0 (0) | 0 (0) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Drafts of any and all publications or presentations of this study must be submitted at least 30 days prior to submission for publication or presentation to Pearl Therapeutics for review, approval, and to ensure consistency. Pearl Therapeutics has the right to request appropriate modification to correct facts and to represent its opinions, or the opinions of the publication committee, if these differ with the proposed publication.